CLINICAL TRIAL: NCT05805631
Title: Efficacy of Intrathecal Pemetrexed Combined With Tyrosine Kinase Inhibitor for Treating Leptomeningeal Metastasis in EGFR-Mutant NSCLC After Failure of Osimertinib
Brief Title: Intrathecal Pemetrexed for Leptomeningeal Metastasis in EGFR-Mutant NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-12-005C
Record Dates: First submitted 2023-03-14; First posted 2023-04-10 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Epidermal Growth Factor Receptor; Leptomeningeal Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Intrathecal pemetrexed combined with EGFR-TKI (physician choice)
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Intrathecal Pemetrexed

SUMMARY:
Leptomeningeal metastasis (LM) is a complication of advanced non-small cell lung cancer (NSCLC). The incidence of LM in NSCLC patients is around 3-5 %, reaching 9.4 % of those with an epidermal growth factor receptor (EGFR) mutation. Generally, the efficacy of systemic treatment for LM is limited due to the blood-brain barrier. Osimertinib has a high central nervous system penetration rate, making it the preferred first-line treatment for EGFR-mutant NSCLC. Previous studies indicated that osimertinib had shown promising efficacy in pretreated patients harboring EGFR mutations and LM. However, intracranial disease progression eventually develops, and the prognosis of patients with LM progression after osimertinib is poor. Recently, intrathecal chemotherapy with pemetrexed (IP) was reported to be an alternative treatment in patients with NSCLC and LM. The results from a phase I/II trial examining the efficacy and safety of IP in patients with EGFR-mutant NSCLC after the failure of previous TKI, and 83% of study enrollees received osimertinib before IP. The clinical response rate was 84.6%, and the median overall survival was 9.0 months. Despite initial promising efficacy, further trials are needed to verify these results. Therefore, the investigators plan to conduct a prospective study to examine the safety and effectiveness of IP combined with EGFR-TKI for patients with EGFR mutant NSCLC after osimertinib failure.

DETAILED DESCRIPTION:
Leptomeningeal metastasis (LM) is a complication of advanced non-small cell lung cancer (NSCLC). The incidence of LMC in NSCLC patients is around 3-5 %, and reaches 9.4 % of those with an epidermal growth factor receptor (EGFR) mutation. Although EGFR tyrosine kinase inhibitors (TKIs) had markedly prolonged survival in advanced NSCLC patients, the prognosis of patients with LMC remains poor. In a Taiwanese NSCLC cohort, the median survival of patients after diagnosis of LMC was 4.5 months. The diagnosis of LM is difficult, and depends on clinical, CSF, and radiographic findings. A positive cerebrospinal fluid (CSF) cytology remains the gold standard for the diagnosis of LM, but the sensitivity of initial lumbar puncture has been reported to be as low as 50%. A gadolinium-enhanced MRI of brain and spine is the best imaging technique for the diagnosis of LM. In patients with metastatic NSCLC and typical presentations of LM, the typical abnormal enhancement on MRI alone can lead to the diagnosis of LMC. However, 20-30% of patients with LM have a normal or false negative MRI. The current diagnostic algorism is based on EANO-ESMO guideline including clinical findings, neuroimaging features and CSF analysis.

The management of LM in patients with NSCLC remained questioned. The aim of treatment is palliative, including amelioration of neurological symptoms, improvement of quality of life, and prolongation of survival. Generally, the efficacy of systemic treatment is limited due to blood-brain barrier. A retrospective study suggests that patients who received contemporary systemic treatment had a decreased risk of death compared to those who did not receive modern systemic therapy. The role of local radiotherapy, in the other hand, is to ease symptoms, to reduce bulky or nodular disease, and to correct CSF flow. There is no consensus on whether whole-brain radiotherapy is a beneficial treatment for patients with leptomeningeal metastasis from NSCLC. Other managements includes intrathecal chemotherapy, CSF diversion surgery, immunotherapy and palliative care.

Osimertinib, a third-generation EGFR-TKI targeting both EGFR sensitizing and T790M resistance mutations, prolonged survival in patients with NSCLC with T790M mutation after EGFR-TKI failure. Compared with other EGFR-TKIs, osimertinib has a high central nervous system (CNS) penetration rate, making it the preferred first-line treatment for EGFR-mutant NSCLC. Previous studies indicated that osimertinib had shown promising efficacy in pretreated patients with EGFR T790M mutation and LM. However, intracranial disease progression eventually develops and the prognosis of patients with LM progression after osimertinib is poor, with a median survival of 7.2 months. Dose intensification of osimertinib to 160 mg per day is a treatment option in patients with EGFR mutant NSCLC and LM after osimertinib failure. In a phase II study by Park et al., patients with T790M-positive NSCLC with brain metastasis and LM were treated with osimertinib 160 mg. Their median PFS and OS were 8.0 and 13.3 months, respectively. A total of 42 percent of patients in the LM cohort received prior T790M targeted agents (osimertinib: 12.5%), and the intracranial disease control rate was 88.2%. In the LM cohort, PFS was not significantly different between patients who had received prior T790M targeted agents and those who did not. In a retrospective study in United States, the median duration of CNS control in patients who received high dose osimertinib was 6.0 months in isolated leptomeningeal progression. The most common adverse events were decreased appetite, diarrhea, and skin rash; however, most were mild in the previous study. More treatment options were needed in this group of patients.

Pemetrexed in a standard chemotherapy regimen in patients with advanced non-squamous NSCLC and showed efficacy in patients with symptomatic brain metastasis. Recently, intrathecal chemotherapy with pemetrexed was reported to be an alternative treatment in patients with NSCLC and LM. In a pilot phase 1 study in China, Pan et al. enrolled thirteen patients and found that maximally tolerated dose of intrathecal pemetrexed (IP) was 10 mg. Severe adverse events were noted in 31% (4/13) of the cases, including myelosuppression, radiculitis, and elevation of hepatic aminotransferases. Another case report also showed a good treatment response to IP (30mg) via Ommaya reservoir in a patient with EGFR mutant NSCLC and LM. Furthermore, Fan et al. published the results from a phase I/II trial examining the efficacy and safety of IP in patients with EGFR mutant NSCLC after failure of previous TKI, and 83% of study enrollees received osimertinib before intrathecal pemetrexed. The clinical response rate was 84.6% and the median overall survival was 9.0 months. The recommended dose of IP was 50 mg with few adverse effects. Despite initial promising efficacy, further trials are need to verify the results.

Therefore, the investigators plan to conduct a prosepctive study to exam the safety and efficacy of IP combined with EGFR-TKI for patients with EGFR mutant NSCLC after osimertinib failure.

ELIGIBILITY:
Inclusion criteria

* At least 20 years of age.
* Patients with metastatic non-squamous NSCLC harboring known EGFR activating mutation and with a diagnosis of probable or confirmed LM by the European Association of Neuro-Oncology-European Society for Medical Oncology (EANO-ESMO) guideline. [5] EGFR activating mutations include exon19 deletion, T790M, L858R, G719X, L861Q, or S768I.
* Intracranial disease progression after osimertinib use, proved by contrast-enhanced MRI
* Stable extra-cranial disease status, judged by investigators.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3 and a minimum life expectancy of 12 weeks
* Normal bone marrow and organ function as defined below:

  * Marrow: Hemoglobin ≥9gm/dL, ANC ≥1500/mm3 platelets ≥100,000/mm3
  * Hepatic: Serum total bilirubin ≤1.5 x upper limit of normal (ULN), ALT (SGPT) and AST (SGOT) ≤3 x ULN.
  * Renal: Creatinine clearance (Ccr) ≥45 mL/min.
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of IP. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* Ability to understand and willingness to sign an IRB approved written informed consent document.
* Willing to provide CSF and plasma samples for ctDNA analysis.

Exclusion criteria

* Uncontrolled extra-CNS disease which needs other systemic treatment than EGFR-TKI.
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN). Patients who are receiving denosumab prior to study enrollment must be willing and eligible to receive a bisphosphonate instead while in the study.
* Malignancies other than NSCLC within 5 years prior to study enrollment, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* On chronic systemic steroid therapy more than 20 mg prednisolone per day (or equivalent) or on any other form of immunosuppressive medication
* Has received a live-virus vaccination within 30 days of planned treatment start
* Systemic cytotoxic chemotherapy or major surgery within 2 weeks of the first dose of study medication
* Active infection requiring therapy
* History of Human Immunodeficiency Virus (HIV) infection.
* Hepatitis B carrier: Patients with HBV infection were required to be receiving effective antiviral therapy and have a viral load less than 100 IU/mL at screening
* Active Hepatitis C
* Has received intrathecal chemotherapy within 2 weeks before the start of IP
* Has received whole-brain radiotherapy (WBRT) within 2 weeks before the start of IP
* Uncontrolled epilepsy
* History of allergic reaction to intravenous pemetrexed.
* Severe coagulation abnormality (INR > 2).
* Severe symptomatic hydrocephalus that requires other treatment modalities other than IP
* Bulky intra-cranial lesion that requires other treatment modalities other than IP

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | Every 6 weeks till disease progression, an average of 6 months
  The response to treatment was determined by combining neurological examination, CSF cytology, and radiographic evaluation by RANO-LM proposal.

SECONDARY OUTCOMES:
Progression-free Survival, LM (PFS-LM) | Every 6 weeks till disease progression, an average of 6 months
  PFS is measured from the date of study enrollment to documented progression of LM according to RANO LM working group or death from any cause.
Progression-free Survival (PFS) | Every 3 months till disease progression, an average of 6 months
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Overall survival (OS) | Every 3 months through study completion , an average of 12 months
  OS is measured from date of study enrollment to the date of death from any cause

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan